CLINICAL TRIAL: NCT03080090
Title: YMCA Exercise Intervention for Smoking Cessation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); YMCA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12-0049
Record Dates: First submitted 2017-02-24; First posted 2017-03-15 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Exercise (Experimental): Individuals in this condition will engage in aerobic exercise 3 times a week for 25 minutes each at 60% to 85% of age-predicted HRmax and smoking cessation intervention through a national quitline while using nicotine replacement patches.
  Interventions: Behavioral: Aerobic exercise; Behavioral: Smoking Cessation Intervention
- Low Intensity Exercise (Active Comparator): The intervention procedures for this group are identical to the Experimental Group group except that the target training intensity will be low intensity exercise, self-selected at 20% to 40% of age-predicted HRmax.
  Interventions: Behavioral: Aerobic exercise; Behavioral: Smoking Cessation Intervention

INTERVENTIONS:
Behavioral: Aerobic exercise — Individuals will work with a YMCA personal trainer to engage in aerobic exercise 3 times a week (25 mins each) for 15 weeks.
Behavioral: Smoking Cessation Intervention — Individuals will work with a national quitline to help them with their smoking cessation goals and make a quit attempt at week 5 of the program.

SUMMARY:
Cigarette smoking is the leading cause of death and disability in the United States. Although smoking has declined since 1964, it is still very common among some groups of people. One such group is persons with emotional symptoms and disorders. There has been little success in developing treatments for smoking cessation for smokers with affective disturbances.

Recent work suggests that being sensitive to, and less tolerant of, stress is associated with many problems in daily life. People with high 'stress sensitivity' tend to use avoidant strategies to cope with their stress, like smoking. Also, people with high levels of stress sensitivity report stronger beliefs that smoking will reduce negative feelings. They also report having a harder time quitting and in fact, are less successful at doing so. This information suggests that stress sensitivity is important to target during smoking cessation treatment for smokers with affective vulnerabilities.

This clinical trial will evaluate a treatment that integrates exercise to reduce stress sensitivity among high stress sensitive smokers. It builds directly from our recent work and we now seek to adapt it to a more a more accessible and sustainable application. Results will provide important information on the benefit of an integrated intervention that could be used in the community for smokers at great risk for relapse and who do not benefit from existing alternative treatments. This study is the first to test an intervention for stress sensitive smokers and has the potential to help at-risk individuals experience quitting success and, ultimately, reduce the burden of tobacco-related cancers in Texas.

DETAILED DESCRIPTION:
Experimental Group. Participants will select a YMCA branch and be assigned a personal fitness instructor who will act as their case manager, overseeing the integrated exercise-based intervention for smoking cessation. Guided by our pilot data showing efficacy and tolerability of the exercise dose, the exercise intervention consists of 75 minutes/week of aerobic training at vigorous-intensity for 15 weeks2. As in the previous study, the aerobic training component will be completed on a treadmill and target training intensity will be self-selected at 60% to 85% of age-predicted heart rate reserve (i.e., vigorous intensity) 2. In order to maximize adherence, the days of the week and training progression schedule will be individualized for each participant based on initial fitness level, travel, and any other issues.

The participant and fitness instructor will meet for three sessions during the first week of exercise training. During the first session, the fitness instructor will describe the program (i.e., treatment model and aims), set a target quit attempt for week 6, develop an exercise training schedule, and supervise the first exercise session to ensure the participant is exercising properly. After two more supervised exercise sessions during the first week, the pair will meet one day per week during the following 14 weeks of the study. The fitness instructors will be responsible for monitoring sessions weekly, problem-solving any difficulties, adjusting the aerobic and/or resistance training regimen as appropriate, and entering the participants exercise data into the (REDCap) database specifically designed for the study.

At the beginning of week 3, the fitness instructor will connect the participant with the quitline (i.e., warm transfer). The Tobacco quitlines are now available in every U.S. state via a national quitline portal, 1-800-QUIT-NOW, and have become the major vehicle through which smoking cessation services are delivered in the U.S.73. All participants will receive the standard telephone counseling package of up to 5 proactive calls from the Texas Tobacco Quitline (https://www.quitnow.net/texas/); we will use a 'warm transfer' (i.e., call the quitline in the presence of the smoker and put them on the phone for the intake interview). Call 1 is an assessment and planning call, Call 2 is a pre-quit date call, Call 3 is a quit date call, and Calls 4 and 5 are maintenance calls if the smoker has quit or problem solving calls if they have not quit. Overall, the counseling protocol aims to (1) provide cognitive-behavioral smoking cessation and relapse prevention tools, tailored to the individual smoker's characteristics and; (2) provide medication management and advice regarding nicotine patch use and adherence support, with the goal of completing a full course of medication - in this case, 8 weeks of transdermal nicotine patch use.

On the target quit day, the fitness instructor will provide the participants with Nicoderm CQ®, 24-hour transdermal nicotine patches (TNP) as part of the study. We chose to provide the patch for 8 weeks because longer than 8 weeks does not appear to improve treatment efficacy10. We chose the TNP because of the extensive empirical literature supporting its effectiveness and safety, its ease of use, and its relatively benign side effect profile that have led to its approval as an over-the-counter medication74. Quitline staff provide instructions on dose and tapering schedule in a fashion consistent with that used in previous trials with a similar formulation of the patch10.

Control Group. The intervention procedures for this group are identical to the Experimental Group group except that the target training intensity will be self-selected at 20% to 40% of age-predicted heart rate reserve (i.e., light intensity).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ages 18-65
* Willing and able to provide informed consent, attend all study visits and comply with the protocol
* Daily smoker for at least one year
* Currently smoke an average of at least 5 cigarettes per day
* Report a motivation to quit smoking in the next month of at least 5 on a 10-point scale.
* Anxiety Sensitivity Index-3 score ≥ 23 (cut-off score to identify high AS individuals)
* Sedentary as defined by moderate-intensity exercise less than 3 days/wk for at least 20 minutes each time
* Medical clearance to participate in the protocol

Exclusion Criteria:

* Use of other tobacco products (including e-cigarettes)
* A lifetime history of bipolar disorder, schizophrenia, psychosis, or delusional disorders; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
* Patients with significant suicidal ideation as determined by structured interview or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Body mass index 40. We selected a BMI of 39.9 as the upper limit in order to screen out individuals with Class III obesity who might be more prone to musculoskeletal injuries than individuals with a BMI<40.0).
* Current use of any psychotherapy for smoking cessation not provided by the researchers.
* Current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers during the quit attempt, including Chantix, Zyban, and Nicotine Replacement Treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Smoking Status after Quit Attempt | 6 weeks
  Change from baseline in point prevalence abstinence (PPA) after quit attempt at week 6 of the protocol.
Smoking Status 1 Month after Quit Attempt | Week 10
  Change from baseline in point prevalence abstinence (PPA) after quit attempt at week 10 of the protocol.
Smoking Status 2 Months after Quit Attempt | Week 14
  Change from baseline in point prevalence abstinence (PPA) after quit attempt at week 14 of the protocol.
Smoking Status 3 Months after Quit Attempt | Week 18
  Change from baseline in point prevalence abstinence (PPA) after quit attempt at week 18 of the protocol.
Smoking Status 6 Months after Quit Attempt | Week 30
  Change from baseline in point prevalence abstinence (PPA) after quit attempt at week 30 of the protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smits JAJ, Rinck M, Rosenfield D, Beevers CG, Brown RA, Conroy Busch HE, Dutcher CD, Perrone A, Zvolensky MJ, Garey L. Approach bias retraining to augment smoking cessation: A pilot randomized controlled trial. Drug Alcohol Depend. 2022 Sep 1;238:109579. doi: 10.1016/j.drugalcdep.2022.109579. Epub 2022 Jul 25. PMID 35917763
- [Derived] Smits JAJ, Zvolensky MJ, Rosenfield D, Brown RA, Otto MW, Dutcher CD, Papini S, Freeman SZ, DiVita A, Perrone A, Garey L. Community-based smoking cessation treatment for adults with high anxiety sensitivity: a randomized clinical trial. Addiction. 2021 Nov;116(11):3188-3197. doi: 10.1111/add.15586. Epub 2021 Jun 13. PMID 34033178